CLINICAL TRIAL: NCT07237126
Title: Efficacy and Safety Assessment of Single-port Robotic Radical Gastrectomy for Gastric Cancer: a Phase 2a Trial Based on the IDEAL Framework
Brief Title: Single-port Robotic Radical Gastrectomy for Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPORTS-04
Record Dates: First submitted 2025-11-16; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer Patients Undergoing Gastrectomy
Keywords: Single-port robotic; Gastric cancer; Radical Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-port Robotic Radical Gastrectomy for Gastric Cancer (Experimental): Single-port Robotic Radical Gastrectomy for Gastric Cancer
  Interventions: Procedure: Single-port Robotic Radical Gastrectomy for Gastric Cancer

INTERVENTIONS:
Procedure: Single-port Robotic Radical Gastrectomy for Gastric Cancer — Single-port Robotic Radical Gastrectomy for Gastric Cancer

SUMMARY:
This study is a single-center, phase 2a exploratory clinical study based on IDEAL framework. The intraoperative and postoperative complications were analyzed to evaluate the safety, feasibility and clinical efficacy of single-port robot-assisted gastric tumor resection.

DETAILED DESCRIPTION:
The study assessed the intraoperative adverse events (device-related and/or procedure-related), postoperative complications, perioperative recovery outcomes, surgical specimen quality, and pathological indices of Single-port robot-assisted radical gastrectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age: 18-75 years; (2) Histologically confirmed gastric adenocarcinoma by endoscopic biopsy; (3) Preoperatively staged as either endoscopically unresectable T1, or cT2-4a with or without nodal involvement (N-/+), and no distant metastasis (M0), according to the 7th edition of the AJCC Cancer Staging Manual; (4) Eligible for potentially curative surgical resection; (5) Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1; (6) American Society of Anesthesiologists (ASA) physical status classification of I-III; (7) Provision of written informed consent.

Exclusion Criteria:

* (1) Pregnant or lactating women; (2) Severe psychiatric disorder; (3) History of prior upper abdominal surgery; (4) Previous gastrectomy, endoscopic submucosal dissection (ESD), or endoscopic mucosal resection (EMR); (5) Preoperative imaging showing regional lymphadenopathy with lymph node(s) larger than 3 cm in diameter; (6) History of another primary malignancy within the past 5 years; (7) Prior neoadjuvant chemotherapy or radiotherapy; (8) History of cerebrovascular or cardiovascular event (e.g., stroke or myocardial infarction) within the past 6 months; (9) Systemic corticosteroid use for more than one month within the past month; (10) Requirement for concomitant surgery for other conditions; (11) Need for emergency surgery due to gastric cancer-related complications (e.g., bleeding, obstruction, or perforation); (12) Participation in another interventional clinical trial previously; (13) Active severe infectious disease; (14) Severe systemic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Intraoperative adverse events and 30-day postoperative complications | Intraoperative and postoperative 30 days
  Intraoperative adverse events (device and/or procedure-related). Events were recorded as Preferred Term and classified under System Organ Class as per MedDRA Common Terminology Criteria for Adverse Events (CTCAE) coding guidelines (https://evs.nci.nih.gov/ftp1/CTCAE/About.html). Postoperative complications will refer to any medical occurrence directly attributed to the surgical procedure within the first 30 days.
Conversion rate | Intraoperative
  Conversion to open or laparotomy surgery due to intraoperative complications , technical difficulties, or inability to successfully complete predefined procedural steps .

SECONDARY OUTCOMES:
Length of incision | Intraoperative
  The total length (in centimeters) of the surgical skin incision made during the procedure, measured immediately after wound closure.
Intraoperative Blood Loss | Intraoperative
  The estimated volume of blood lost during surgery (in milliliters), calculated based on suction collection volume and the weight of used gauze sponges, using standard conversion methods.
Operative Time | Intraoperative
  The duration (in minutes) from the initial skin incision to final wound closure, excluding anesthesia induction and emergence.
Postoperative Length of Hospital Stay | 7 days after surgery
  The number of days between the day of surgery (postoperative day 0) and the day of hospital discharge, inclusive of the discharge day if applicable per institutional protocol.
Number of Lymph Nodes Harvested | 7 days after surgery
  The total count of lymph nodes removed during the lymphadenectomy and confirmed by pathological examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ito A, Nakauchi M, Fujita M, Umeki Y, Suzuki K, Serizawa A, Akimoto S, Watanabe Y, Tanaka T, Shibasaki S, Inaba K, Uyama I, Suda K. Initial clinical experiences of robotic distal gastrectomy for gastric cancer using the Da Vinci SP system: a single-center retrospective study. Langenbecks Arch Surg. 2025 Mar 29;410(1):110. doi: 10.1007/s00423-025-03685-w. PMID 40156763
- [Background] Park SH, Kim YN, Hwang J, Kim KY, Cho M, Kim YM, Hyung WJ, Kim HI. Safety and feasibility of reduced-port robotic distal gastrectomy for gastric cancer: a phase I/II clinical trial using the da Vinci Single Port(SP) robotic system. Sci Rep. 2023 Oct 30;13(1):18578. doi: 10.1038/s41598-023-45655-6. PMID 37903856
- [Background] Shang L, Zhang R, Dong K, Xiao K, Zheng C, Shi Y, Liu H, Jing C, Li L. The world's first pure single-port robotic radical total gastrectomy for advanced gastric cancer. Chin Med J (Engl). 2024 Dec 20;137(24):3151-3152. doi: 10.1097/CM9.0000000000003380. Epub 2024 Nov 28. No abstract available. PMID 39604102
- [Background] Qiu WW, Huang ZN, Li TY, Zhang L, She JJ, Jia BQ, Qin XG, Ren SY, Yao HL, Liu DN, Liang H, Shi FY, Li P, Li BP, Zhang XS, Liu KJ, Zheng CH, Lin JX, Huang CM, Li P. Comparison of short- and mid-term outcomes of robotic versus laparoscopic gastrectomy in high-risk patients with gastric cancer: a nationwide, multicentre cohort study. Eur J Surg Oncol. 2025 Oct;51(10):110294. doi: 10.1016/j.ejso.2025.110294. Epub 2025 Jul 3. PMID 40651456
- [Background] Keller DS, Reif de Paula T, Ikner TP, Saidi H, Schoonyoung H, H Marks J. Perioperative outcomes for single-port robotic versus single-incision laparoscopic surgery: a comparative analysis in colorectal cancer surgery. Surg Endosc. 2024 Mar;38(3):1568-1575. doi: 10.1007/s00464-023-10629-2. Epub 2024 Jan 4. PMID 38177611
- [Background] Cheng X, Huang C, Jia W, Guo Z, Shi Y, Song Z, Feng H, Huang H, Xu S, Li H, Wang S, Zhang Y, Zhang T, Liu K, Ji X, Zhao R. Clinical status and future prospects of single-incision robotic-assisted surgery: a review. Int J Surg. 2023 Dec 1;109(12):4221-4237. doi: 10.1097/JS9.0000000000000944. PMID 37988410
- [Background] Cianchi F, Staderini F, Badii B. Single-incision laparoscopic colorectal surgery for cancer: state of art. World J Gastroenterol. 2014 May 28;20(20):6073-80. doi: 10.3748/wjg.v20.i20.6073. PMID 24876729
- [Background] Markar SR, Karthikesalingam A, Di Franco F, Harris AM. Systematic review and meta-analysis of single-incision versus conventional multiport appendicectomy. Br J Surg. 2013 Dec;100(13):1709-18. doi: 10.1002/bjs.9296. PMID 24227355
- [Background] Haueter R, Schutz T, Raptis DA, Clavien PA, Zuber M. Meta-analysis of single-port versus conventional laparoscopic cholecystectomy comparing body image and cosmesis. Br J Surg. 2017 Aug;104(9):1141-1159. doi: 10.1002/bjs.10574. Epub 2017 Jun 1. PMID 28569406
- [Background] Seo HS, Lee HH. Is the 5-ports approach necessary in laparoscopic gastrectomy? Feasibility of reduced-port totally laparoscopic gastrectomy for the treatment of gastric cancer: A Prospective Cohort Study. Int J Surg. 2016 May;29:118-22. doi: 10.1016/j.ijsu.2016.03.035. Epub 2016 Mar 28. PMID 27034118
- [Background] Liu Y, Yun H, Zhang W, Zou H, Chen N, Wang Y, Luo Z, Xu X, Sun Y, Chen Y, Beznosenko A, ALMasri H, McClure MA, Ma H, Yu J, Lv Q. Robotic versus laparoscopic total gastrectomy for gastric cancer: a systematic review and meta-analysis of perioperative and oncologic outcomes. Int J Surg. 2025 Sep 1;111(9):6397-6411. doi: 10.1097/JS9.0000000000002761. Epub 2025 Jun 19. PMID 40549444
- [Background] Li Z, Zhou W, Yang W, Miao Y, Zhang Y, Duan L, Niu L, Chen J, Fan A, Xie Q, Wei S, Bai H, Wang C, Chen X, Han Y, Hong L. Efficacy and safety of robotic vs. laparoscopic gastrectomy for patients with gastric cancer: systematic review and meta-analysis. Int J Surg. 2024 Dec 1;110(12):8045-8056. doi: 10.1097/JS9.0000000000001826. PMID 38874467
- [Background] Jayne D, Pigazzi A, Marshall H, Croft J, Corrigan N, Copeland J, Quirke P, West N, Rautio T, Thomassen N, Tilney H, Gudgeon M, Bianchi PP, Edlin R, Hulme C, Brown J. Effect of Robotic-Assisted vs Conventional Laparoscopic Surgery on Risk of Conversion to Open Laparotomy Among Patients Undergoing Resection for Rectal Cancer: The ROLARR Randomized Clinical Trial. JAMA. 2017 Oct 24;318(16):1569-1580. doi: 10.1001/jama.2017.7219. PMID 29067426
- [Background] Kim HH, Han SU, Kim MC, Kim W, Lee HJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Hyung WJ; Korean Laparoendoscopic Gastrointestinal Surgery Study (KLASS) Group. Effect of Laparoscopic Distal Gastrectomy vs Open Distal Gastrectomy on Long-term Survival Among Patients With Stage I Gastric Cancer: The KLASS-01 Randomized Clinical Trial. JAMA Oncol. 2019 Apr 1;5(4):506-513. doi: 10.1001/jamaoncol.2018.6727. PMID 30730546
- [Background] Katai H, Mizusawa J, Katayama H, Morita S, Yamada T, Bando E, Ito S, Takagi M, Takagane A, Teshima S, Koeda K, Nunobe S, Yoshikawa T, Terashima M, Sasako M. Survival outcomes after laparoscopy-assisted distal gastrectomy versus open distal gastrectomy with nodal dissection for clinical stage IA or IB gastric cancer (JCOG0912): a multicentre, non-inferiority, phase 3 randomised controlled trial. Lancet Gastroenterol Hepatol. 2020 Feb;5(2):142-151. doi: 10.1016/S2468-1253(19)30332-2. Epub 2019 Nov 19. PMID 31757656
- [Background] Hyung WJ, Yang HK, Park YK, Lee HJ, An JY, Kim W, Kim HI, Kim HH, Ryu SW, Hur H, Kim MC, Kong SH, Cho GS, Kim JJ, Park DJ, Ryu KW, Kim YW, Kim JW, Lee JH, Han SU; Korean Laparoendoscopic Gastrointestinal Surgery Study Group. Long-Term Outcomes of Laparoscopic Distal Gastrectomy for Locally Advanced Gastric Cancer: The KLASS-02-RCT Randomized Clinical Trial. J Clin Oncol. 2020 Oct 1;38(28):3304-3313. doi: 10.1200/JCO.20.01210. Epub 2020 Aug 20. PMID 32816629
- [Background] Wang FH, Zhang XT, Tang L, Wu Q, Cai MY, Li YF, Qu XJ, Qiu H, Zhang YJ, Ying JE, Zhang J, Sun LY, Lin RB, Wang C, Liu H, Qiu MZ, Guan WL, Rao SX, Ji JF, Xin Y, Sheng WQ, Xu HM, Zhou ZW, Zhou AP, Jin J, Yuan XL, Bi F, Liu TS, Liang H, Zhang YQ, Li GX, Liang J, Liu BR, Shen L, Li J, Xu RH. The Chinese Society of Clinical Oncology (CSCO): Clinical guidelines for the diagnosis and treatment of gastric cancer, 2023. Cancer Commun (Lond). 2024 Jan;44(1):127-172. doi: 10.1002/cac2.12516. Epub 2023 Dec 31. PMID 38160327
- [Background] Sun D, Mulder DT, Li Y, Nieboer D, Park JY, Suh M, Hamashima C, Han W, O'Mahony JF, Lansdorp-Vogelaar I. The Effect of Nationwide Organized Cancer Screening Programs on Gastric Cancer Mortality: A Synthetic Control Study. Gastroenterology. 2024 Mar;166(3):503-514. doi: 10.1053/j.gastro.2023.11.286. Epub 2023 Nov 24. PMID 38007053
- [Background] Chen Y, Jia K, Xie Y, Yuan J, Liu D, Jiang L, Peng H, Zhong J, Li J, Zhang X, Shen L. The current landscape of gastric cancer and gastroesophageal junction cancer diagnosis and treatment in China: a comprehensive nationwide cohort analysis. J Hematol Oncol. 2025 Apr 15;18(1):42. doi: 10.1186/s13045-025-01698-y. PMID 40234884
- [Background] Yang WJ, Zhao HP, Yu Y, Wang JH, Guo L, Liu JY, Pu J, Lv J. Updates on global epidemiology, risk and prognostic factors of gastric cancer. World J Gastroenterol. 2023 Apr 28;29(16):2452-2468. doi: 10.3748/wjg.v29.i16.2452. PMID 37179585
- [Background] Park JY, Georges D, Alberts CJ, Bray F, Clifford G, Baussano I. Global lifetime estimates of expected and preventable gastric cancers across 185 countries. Nat Med. 2025 Sep;31(9):3020-3027. doi: 10.1038/s41591-025-03793-6. Epub 2025 Jul 7. PMID 40624406